CLINICAL TRIAL: NCT03828604
Title: Stress-Induced Inflammation and Reward Processing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Chloe Boyle, PhD, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SIWB
Record Dates: First submitted 2019-01-31; First posted 2019-02-04 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Stress, Psychological
Keywords: reward processing
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Acute Psychosocial stress vs. Non-stress active control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress; Trier Social Stress Task (Experimental): 5 min challenging speech task, 5 min challenging math task; performed in front of evaluators
  Interventions: Behavioral: Stress; Trier Social Stress Task
- Placebo Trier Social Stress Task (Active Comparator): 5 min speech task, 5 min math task; performed alone
  Interventions: Behavioral: Placebo Trier Social Stress Task

INTERVENTIONS:
Behavioral: Stress; Trier Social Stress Task — Standardized acute psychosocial stressor
  Arms: Stress; Trier Social Stress Task
Behavioral: Placebo Trier Social Stress Task — Active control version of the TSST
  Arms: Placebo Trier Social Stress Task

SUMMARY:
Anhedonia, or loss of interest or pleasure, is a key feature of depression and transdiagnostic construct in psychopathology. Both theory and compelling evidence from preclinical models implicates stress-induced inflammation as a key psychobiological pathway to anhedonic behavior; however, this pathway has not been demonstrated in human models. Further, although anhedonia may reflect dysregulation in multiple dimensions of reward, the extent to which stress-induced inflammation alters these dimensions is unclear. The current placebo controlled study used a standardized laboratory stressor task to elicit an inflammatory response in a sample of a healthy young women and evaluate effects of stress-induced inflammation on multiple behavioral indices of reward processing.

DETAILED DESCRIPTION:
In this study we propose to examine the association between psychosocial stress, the stress-induced inflammatory response, and reward processing in a female undergraduate sample. Specifically, we will 1) examine effects of an acute psychosocial stressor on reward processing; 2) evaluate the association between stress-related changes in inflammation and reward processing; and 3) test key vulnerability factors that may moderate the association between stress and reward. To achieve these goals, this study will recruit 60 female undergraduate students to test effects of stress on reward processing in a 3.5 hour laboratory session. Participants will be randomly assigned to either experience a laboratory stressor or a placebo control, and will complete reward tasks 90 minutes post stress/placebo onset, at which point the peripheral inflammatory response to stress reaches its peak. The reward tasks are computerized behavioral tasks that assess three domains of reward processing: reward-learning, reward motivation, and reward sensitivity. Throughout the session, all participants will complete self-report measures of affect and provide blood and saliva samples for evaluation of the psychological and physiological stress response. Within one week prior to the session, participants will attend a 1 hour visit in which they complete baseline reward tasks and self-report questionnaires assessing mood, personality, early life stress, and health behaviors. In total, participants will complete two visits, with a duration of 4.5 hours. This study builds upon prior studies demonstrating immediate effects of acute stress on reward processing, and further tests for delayed effects of acute stress on reward processing. Furthermore, this will be the first study to examine inflammation as a mechanism linking stress to deficits in reward processing. Findings may inform theory of depression etiology and contribute to more specialized treatment that is targeted at specific symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* English fluency
* Age 18-28
* Biologically female

Exclusion Criteria:

* Current illness
* Presence or history of major medical conditions
* Current or past diagnosis of alcohol use disorder
* Use of tobacco
* Use of immune-altering medications
* Current pregnancy

Ages: 18 Years to 28 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 57 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2018-05-09 (Actual)

PRIMARY OUTCOMES:
Probabilistic Reward Task - Reward Responsiveness | Pre-TSST/P-TSST and 90 min post-TSST/P-TSST
  Change in the magnitude of response bias from pre to post Trier Social Stress Task (TSST) or Placebo-TSST (P-TSST).
Effort Expenditure for Rewards Task - Reward Motivation | Pre-TSST/P-TSST and 120 min post-TSST/P-TSST
  Change in amount of hard trials chosen from pre to post-TSST/P-TSST (overall, and at 3 levels of probability of potential rewards; low, medium, and high)
Attentional Bias Task | Pre-TSST/P-TSST and 110 min post-TSST/P-TSST
  Change in attentional bias from pre to post-TSST/P-TSST

SECONDARY OUTCOMES:
Effort Expenditure for Rewards Task - Reward Sensitivity | 120 min post-TSST
  Strength of the relationship between changes in reward magnitude and high effort trial choice as a function of degree of change in IL-6 following acute stress
Face Morphing Task | Pre-TSST/P-TSST and 115 min post-TSST/P-TSST
  Change in latency to detect emotional expressions

OTHER OUTCOMES:
Depressive symptoms | Change in depressive symptoms from study entry to 4-month follow-up
  The 20-item Center for Epidemiological Studies Depression Scale (CESD) is a self-report measure; participants are asked to rate how often they have experienced depressed feelings, attitudes, and behavioral symptoms during the past week (0 = rarely; 3 = most of the time). The total score range is 0 to 60, with higher scores indicating higher depressive symptoms.
Affective experience during the experimental session | Entry, pre-TSST/P-TSST; during TSST/P-TSST; 60, 90, 120, 150 min post TSST/P-TSST
  Emotional reactivity and recovery from the TSST/P-TSST will be assessed using items from the Positive and Negative Affect Schedule and the Profile of Mood States. Participants rate how they feel "right now (that is, at the present moment) on a 1 (very slightly or not at all) to 5 (extremely) Likert scale. Average scores for subscales are reported, including positive and negative affect (7 items each), fatigue (8 items) vigor (5 items) and confusion (7 items). Participants also use visual analogue scales (VAS) to indicate how stressed, anxious, angry, confident, calm, socially connected and happy they are currently feeling on a 0 (not at all) to 100 (extremely) scale. The VAS are completed alongside the PANAS and three additional times during the TSST/P-TSST.

CONTACTS AND LOCATIONS:
Overall Officials: Chloe C Boyle, PhD, Principal Investigator — University of California, Los Angeles; Julienne E Bower, PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Clinical and Translational Research Center, University of California, Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Derived] Boyle CC, Stanton AL, Eisenberger NI, Seeman TE, Bower JE. Effects of stress-induced inflammation on reward processing in healthy young women. Brain Behav Immun. 2020 Jan;83:126-134. doi: 10.1016/j.bbi.2019.09.023. Epub 2019 Sep 30. PMID 31580931

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-31): https://cdn.clinicaltrials.gov/large-docs/04/NCT03828604/Prot_SAP_000.pdf